CLINICAL TRIAL: NCT06099093
Title: A Pilot Study of 18F-DCFPyL-PSMA PET in Patients Receiving 177Lu-Vipivotide Tetraxetan Therapy for Metastatic Castrate-resistant Prostate Cancer
Brief Title: Pilot of 18F-DCFPyL-PSMA PET in mCRPC Patients Receiving 117Lu-Vipivotide Tetraxetan
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Heather A. Jacene, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-385
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Metastatic Castration-resistant Prostate Carcinoma
Keywords: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Metastatic Castration-resistant Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; 18F-JK-PSMA-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 18F-DCFPYL-PSMA PET (Experimental): Study procedures will be conducted as follows:
  * Baseline screening visit with PSMA-PET/CT scan with Ga-PSMA-11.
  * In-clinic visit with exam and PSMA-PET/CT scan with 18F-DCFPyl per standard institutional procedures.
  * Standard of care therapy.
  * Follow up every 3 months via chart review for 12 months, with the purpose of seeing how participants respond to 177Luvipivotide tetraxetan treatment.
  Interventions: Drug: 18F-DCFPyl

INTERVENTIONS:
Drug: 18F-DCFPyl — Fluorine-labeled small molecule, via intravenous infusion per protocol.
  Other Names: [F18]-Piflufolastat, Pylarify, 2-(3-{1-carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]- pentyl}ureido)-pentanedioic acid

SUMMARY:
The purpose of this research study is to see how well an imaging test, called 18FDCFPyL prostate specific membrane antigen (PSMA) positron emission tomography (PET), can show the extent of prostate cancer when comparing to 68Ga-PSMA-11 PET/CT (another type of diagnostic scan for prostate cancer).

DETAILED DESCRIPTION:
This is a one-arm single-stage prospective pilot study to determine how 18F-DCFPyL PSMA-PET/CT can be used as a diagnostic test before treatment with 177Lu-vipivotide tetraxetan, which is an approved therapy for advanced prostate cancer.

The U.S. Food and Drug Administration (FDA) has approved 18F-DCFPyL as a diagnostic agent (radiotracer) option for prostate cancer, though it is not specifically approved for participants who are due to receive 177Lu-vipivotide tetraxetan therapy.

This research study involves a single PET scan using the imaging agent 18F-DCFPyL and the collection of information from medical records.

Participation in this research study is expected to last about 12 months.

It is expected that about 30 people will take part in this research study. Progenics Pharmaceuticals, Inc. is funding this research study by providing funding and the imaging agent, 18F-DCFPyL.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate cancer.
* Age ≥18 years.
* Participants must be planned for standard-of-care 177Lu-Vipivotide Tetraxetan therapy after the 18F-DCFPyL PSMA-PET.

  -≥1 PSMA-avid lesion on 68Ga-PSMA-11 PSMA-PET performed within 120 days of study entry (to meet eligibility for 177Lu-Vipivotide Tetraxetan therapy).
* Ability and willingness to comply with the study procedures.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational agent are eligible for this trial.
* The effects of 18F-DCFPyL on the developing human fetus are unknown. For this reason and because radiopharmaceutical agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 24 hours after the 18F-DCFPyL PSMA-PET scan.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Contraindications to PET/CT, including severe claustrophobia.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-DCFPyL
* Any past or current condition that, in the opinion of the study investigators, would confound the results of the study or would pose additional risk or burden to the patient by their participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with PSMA-Positive Lesion | 1 Day
  Defined as the number of participants with at least 1 PSMA-positive lesion on 18F-DCFPyL PSMA-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jacene, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu